CLINICAL TRIAL: NCT06962956
Title: An Exploratory Study to Evaluate the Relationship Between Gingivitis and Systemic Biomarkers
Brief Title: Evaluating Gingivitis and Systemic Biomarkers
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2024058
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Negative Control (Active Comparator): 0.76% sodium monofluorophosphate
  Interventions: Drug: 0.76% Sodium Monofluorophosphate Dentifrice
- Test (Active Comparator): 0.454% stannous fluoride
  Interventions: Drug: 0.454% Stannous Fluoride Dentifrice
- Positive Control (Active Comparator): 0.454% stannous fluoride
  Interventions: Drug: 0.454% Stannous Fluoride Dentifrice

INTERVENTIONS:
Drug: 0.76% Sodium Monofluorophosphate Dentifrice — Brush two times a day for 1 minute with manual toothbrush
  Arms: Negative Control
Drug: 0.454% Stannous Fluoride Dentifrice — Brush two times a day for 1 minute with manual toothbrush
  Arms: Test
Drug: 0.454% Stannous Fluoride Dentifrice — Brush two times a day for 2 minutes with electric toothbrush
  Arms: Positive Control

SUMMARY:
This exploratory study will consist of two parts: Phase 1 (sample collection/screening) and Phase 2 (sample collection/product efficacy testing). The purpose of Phase 1 is to understand the association of gingivitis to systemic biomarkers and to screen subjects for Phase 2. The purpose of Phase 2 is to assess the causal effect of oral hygiene intervention on gingivitis and systemic biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent and receive a signed copy of the informed consent form;
* Be between 25 - 65 years of age;
* Have at least 16 gradable teeth;
* Have a minimum of (approximately) 30% of bleeding sites and no more than two teeth with pockets deeper than 5mm or deemed acceptable by the Investigator/Designee (unhealthy test subjects only);
* Have less than or equal to 3 bleeding sites and with all pockets less than or equal to 3mm deep (healthy test subjects only);
* Agree to fast 12 hours prior to any visit with a blood collection;
* Agree to not perform any oral hygiene for at least 12 hours prior to any visit with dental exams, saliva collection, and plaque collections;
* Agree to refrain from eating or drinking, using medicated lozenges, breaths mints, and chewing gum at least 4 hours prior to this study visit (exception allowed: small sips of water up until 45 minutes prior to their appointment) for any visit with plaque collections;
* Agree to refrain from use of any non-study oral hygiene products after the Product Distribution visit;
* Agree to continue their current oral hygiene products and habits until the Product Distribution visit;
* Agree to delay any elective dentistry, including dental prophylaxis outside of the study protocol, until the completion of the study;
* Agree to all study restrictions for the duration of the study (medicines/supplements/vaccines- see restricted list);
* Agree not to participate in any other oral care studies for the duration of this study;
* Agree to return for all scheduled visits and to follow all study procedures; and
* Be in good general health, as determined by the Investigator/Designee based on a review of their health history.

Exclusion Criteria:

* Severe periodontal disease, including but not limited to purulent exudate, generalized mobility, and/or severe recession;
* Active treatment for gingivitis, periodontitis, or caries;
* Daily use of NSAID;
* Having any of the following: fixed orthodontic appliances or attachments for aligner treatment, lower bonded retainers; removable partial dentures, peri/oral piercings, a pacemaker or other implanted device, unless deemed acceptable by the Investigator/Designee;
* A condition requiring the need for antibiotic premedication prior to dental procedures;
* Use of anti-inflammatory or anti-coagulant medications within 2 weeks of the Baseline visit, unless deemed acceptable by the Investigator/Designee;
* Having had oral/gum surgery within the previous 2 months;
* Smoking or vaping (regardless of content), use of smokeless tobacco, e-cigarettes, or nicotine patches);
* Currently using recreational drugs;
* Having been diagnosed with cardiovascular disease, diabetes (having an A1C ≥ 7), rheumatoid arthritis, liver disease, IBS, Crohn's Disease, Chronic Kidney Disease, or any type of autoimmune disease;
* Having any gastrointestinal issues (e.g. diarrhea, vomiting) in the past week;
* Use of statins or cholesterol lowering medication or supplements (e.g., Flax seeds, omega-3 fatty acids, Magnesium Oxide ≥250mg, Zyflamed, supplements containing berberine, golden thread, turmeric, CoQ10, or quercetin) for the duration of the study;
* Use of antibiotics or having a dental prophylaxis in the last 4 weeks prior the baseline visit, unless deemed acceptable by the Investigator/Designee;
* Receiving a flu shot or other vaccination in the last 4 weeks prior the baseline visit;
* Inability to undergo any study procedures;
* Currently undergoing treatment with GLP-1s antagonist;
* Nursing, self-reported pregnancy or the intention of becoming pregnant any time during the course of this study; or
* Having any condition or disease, as determined by the Investigator/Designee based on a review of the medical history which could be expected to interfere with examination procedures or with the subject's safe completion of the study.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Number Bleeding Sites | 4 months
  Total number of bleeding sites

CONTACTS AND LOCATIONS:
Overall Officials: Salus Research, Principal Investigator — Salus Research
Locations (1):
- Salus Research, Fort Wayne, Indiana, United States